CLINICAL TRIAL: NCT03147638
Title: Multi-Center Single Arm Trial to Determine The Effectiveness of Warfarin Therapy Duration For Heparin-Induced Thrombocytopenia (HIT)
Acronym: HIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Yazan Numan, M.D., Marshall University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 943871-5
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — Warfarin; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Intervention Model Description: Single arm with retrospective arm The retrospective arm is he comparator and they are historic control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 month (Experimental): patient treated with Anti coagulation for one month
  Interventions: Drug: Warfarin, NOAC
- 3 months (Active Comparator): standard of care , treatment for 3 months
  Interventions: Drug: Warfarin, NOAC

INTERVENTIONS:
Drug: Warfarin, NOAC — duration of treatment

SUMMARY:
Multi-Center Single Arm Trial to Determine The Effectiveness of Warfarin Therapy Duration For Heparin-Induced Thrombocytopenia (HIT)

ELIGIBILITY:
Inclusion criteria:

* Patient must be able to provide an informed consent
* Patient older than 18 years' old
* Patient with suspected diagnosis of HIT, need 2 of the following:

have a fall in platelet count of > 30% from a baseline prior to heparin/LMWH Platelet factor 4 (PF4) ELISA positive Develop skin lesions secondary to subcutaneous heparin With T score more than 4 For those less than 4 we will use serotonin release assay-SRA

* Patient received the bridging therapy of non-heparin anticoagulant
* Patient is receiving the standard of care treatment for HIT
* Patient is willing to be followed up for by one of the physicians listed in the delegation log
* The Primary physician responsible for the patient is agreeing for the patient to participate
* Patients are not involved in a clinical trial for HIT management

Exclusion Criteria:

* Patient is unable to sign an informed consent
* Patient doesn't have a confirmed diagnosis of HIT
* Patient Does not have Pulmonary embolus
* Patient does is not on Warfarin for other indications
* Patient is a known case of hypercoagulable disorder
* Patient is not willing to come back for follow up
* Patient is critically ill or has a life expectancy of less than 3 months
* Pregnancy that is in First trimester.
* Multi-system organ failure or estimated survival of less than 30 days
* Uncontrolled hypertension defined as a blood pressure >180/110 mm Hg

Ages: 18 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2019-01-11 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
All cause hospitalization | Within six months after treatment
side effects of Warfarin treatment | Within six months after treatment
All cause mortality | Within six months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall University, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No